CLINICAL TRIAL: NCT06525168
Title: Phase I Clinical Study of the Safety, Tolerability, Food Effect and Pharmacokinetics of DA414 Granules After Single and Multiple Administration in Healthy Subjects
Brief Title: Safety, Tolerability and Pharmacokinetic Characteristics Evaluation on DA414
Acronym: DA414
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chendu DIAO Nine Hong Pharmaceutical Factory (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: Chendu DIAO NineHong Factory
Record Dates: First submitted 2024-07-17; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Ischemic Stroke
Keywords: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DA414 Granules (Experimental): The trial plans to conduct studies with five dosage groups. The 12.5 mg dosage group will include 2 subjects, both receiving DA414 granules. The 25 mg, 50 mg, and 100 mg dosage groups will each include 10 subjects randomly assigned in a 8:2 ratio (8 receiving the investigational drug and 2 receiving placebo). The 200 mg dosage group will include 8 subjects, randomly assigned in a 6:2 ratio (6 receiving the investigational drug and 2 receiving placebo).
  Interventions: Drug: DA414 Granules
- DA414 Placebo (Placebo Comparator): The trial plans to conduct studies with five dosage groups. The 12.5 mg dosage group will include 2 subjects, both receiving DA414 granules. The 25 mg, 50 mg, and 100 mg dosage groups will each include 10 subjects randomly assigned in a 8:2 ratio (8 receiving the investigational drug and 2 receiving placebo). The 200 mg dosage group will include 8 subjects, randomly assigned in a 6:2 ratio (6 receiving the investigational drug and 2 receiving placebo).
  Interventions: Drug: DA414 placebo

INTERVENTIONS:
Drug: DA414 Granules — DA414 Granules single ascending doses. DA414 will be orally administrated at single ascending doses of 12.5 mg, 25mg, 50 mg, 100mg and 200 mg.
  Other Names: DA414
  Arms: DA414 Granules
Drug: DA414 placebo — DA414 placebo single ascending doses. DA414 placebowill be orally administrated at single ascending doses of 25mg, 50 mg, 100mg and 200 mg.
  Other Names: Placebo
  Arms: DA414 Placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability, pharmacokinetics (PK) and Food Effects of DA414 Granules in Chinese healthy subjects with single and multiple doses.

DETAILED DESCRIPTION:
Acute ischemic stroke is the most common type of stroke, characterized by high incidence, prevalence, recurrence, disability, and mortality rates, posing a serious threat to public health. However, the current treatment measures are limited and often ineffective. According to existing preclinical data, DA414 has demonstrated significant development potential in both in vitro and in vivo pharmacodynamic studies across multiple batches and models. Based on the data-driven insights, the sponsor will conduct single ascending dose (SAD) studies, multiple ascending dose (MAD) studies, and food effect studies of DA414 in healthy subjects.

ELIGIBILITY:
* Inclusion Criteria:

  1. Subjects are fully aware of the purpose, nature, procedures, and possible adverse effects of the trial, volunteer as subjects, and sign an informed consent form prior to the start of any study procedures;
  2. Healthy subjects aged 18-45 years (including the threshold);
  3. Male weight ≥ 50.0 kg, female weight ≥ 45.0 kg; body mass index (BMI) in the range of 19.0-26.0 kg/m2 (including threshold values);
  4. Subjects are voluntarily using effective contraception during the trial and for 6 months after the last dose, and are not planning to have children or to donate sperm or eggs;
  5. Those who are able to communicate well with the researcher and understand and comply with the requirements of this study.
* Exclusion Criteria:

  1. Have a history of specific allergies (asthma, urticaria, eczema, etc.) or allergic constitution (such as known allergy to two or more substances), or known history of allergy to DA414 and related excipients
  2. Those with an acute illness occurring within 2 weeks prior to screening;
  3. Persons with a history of chronic or serious disease of the cardiovascular, hepatic, renal, biliary, respiratory, hematologic and lymphatic, endocrine, immunologic, psychiatric, neuromuscular, or gastrointestinal systems within one year prior to screening, or a history of gastrointestinal disorders (including existing) within one year prior to screening This includes chronic or active upper gastrointestinal diseases such as esophageal disease, gastritis, duodenitis, peptic ulcers, or active gastrointestinal bleeding, or gastrointestinal surgery;
  4. Screening vital signs, physical examination, clinical laboratory tests (routine blood, urine, blood biochemistry, coagulation, blood transfusion), chest X-ray, abdominal ultrasound (liver, gallbladder, pancreas, spleen and kidneys), and results of clinically significant abnormality as judged by the investigator;
  5. Those whose ECG results showed QTc>440ms at screening (Fridericia's formula correction, calculated as QTcF= QT/(RR0.33));
  6. Those who have undergone major surgical procedures (excluding diagnostic surgical procedures) within 6 months prior to screening, or who are scheduled to undergo surgery during the study period, or who have undergone surgery that, in the judgment of the investigator, would interfere with drug absorption, distribution, metabolism, or excretion;
  7. Those who have used any medications (including any prescription drugs, over-the-counter drugs, herbal preparations and formulas, etc.) and nutraceuticals within 2 weeks prior to the first dose;
  8. Inhibitors or inducers of CYP3A4, CYP2B6 within 30 days prior to first dose e.g., inducers - rifampicin, phenobarbital, carbamazepine, phenytoin; inhibitors - clarithromycin, itraconazole, ketoconazole, ritonavir, azamorelin,zithromycin,verapamil,sertraline, phencyclidine, septiparatide, ticlopidine. azamorelin,zithromycin,verapamil,sertraline, phencyclidine, septiparatide, ticlopidine.
  9. Those who ingested strong tea, caffeine-containing, alcoholic beverages, or foods that interfere with drug metabolism, such as popcorn, papaya, blackberry, grapefruit, or grapefruit products, within 48h prior to drug administration;
  10. Those who had received a live attenuated vaccination within 2 weeks prior to screening or who required live attenuated vaccination during the trial;
  11. Participants who have participated in other clinical trials within 3 months prior to screening (Note: End time is defined as the date of exit from the last clinical trial in which they participated);
  12. Those who have donated blood within 3 months prior to screening, those who have lost a total of 400 mL or more of blood from blood donation or other causes within 6 months (except for normal blood loss during physiological periods in women), or those who have had unexplained abnormal bleeding in the past;
  13. Persons who have consumed an average of more than 2 units of alcohol per week (1 unit = 360 mL of beer or 45 mL of 40% alcohol liquor or 150 mL of wine) during the past year, or who were unable to abstain from alcohol during the test period, or who have had a breath test result of greater than 0.0 mg/100 mL of alcohol;
  14. Those who smoked more than 5 cigarettes per day in the 3 months prior to screening or who were unable to stop using any tobacco products during the trial.
  15. Those with a history of substance abuse (including repeated, heavy non-medical use of all types of narcotic drugs and psychotropic substances) or a positive substance abuse screen (including: morphine, methamphetamine (meth), ketamine, ecstasy (MDMA), marijuana (tetrahydrocannabinolic acid (THC)), etc.) within the past year;
  16. Individuals who cannot tolerate venipuncture/indwelling needles,or who have a history of needle and blood sickness,or who have difficulty swallowing;
  17. lactose-intolerant
  18. Those who have special dietary requirements and cannot accept a uniform diet;
  19. Other subjects judged by the investigator to be unsuitable for participation.Female subjects shall be excluded if, in addition to the above requirements, they meet the following criteria:
  20. Those who used oral contraceptives within 30 days prior to screening;
  21. Use of long-acting estrogen or progestin injections (with progestin-based IUDs) or implants within 6 months prior to screening;
  22. Unprotected sex with partner within 14 days prior to screening
  23. A woman who has a positive pregnancy test or a test result that is not within normal values or within the range of non-pregnant status;
  24. Pregnant or lactating women;

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Estimated)
Dates: Start 2024-02-06 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
safety and tolerability | Through study completion, an average of 28 days.
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0.

SECONDARY OUTCOMES:
Cmax | Measured on 1 hour before administration and 1, 2, 3, 4, 5, 6, 7, 8, 12, 24, 72, 96, 144, 192 hours after administration.
  Plasma samples were collected at different points for pharmacokinetic analysis.
AUC0-t | Measured on 1 hour before administration and 1, 2, 3, 4, 5, 6, 7, 8, 12, 24, 72, 96, 144, 192 hours after administration.
  Plasma samples were collected at different points for pharmacokinetic analysis.
Tmax | Measured on 1 hour before administration and 1, 2, 3, 4, 5, 6, 7, 8, 12, 24, 72, 96, 144, 192 hours after administration.
  Plasma samples were collected at different points for pharmacokinetic analysis.
T1/2 | Measured on 1 hour before administration and 1, 2, 3, 4, 5, 6, 7, 8, 12, 24, 72, 96, 144, 192 hours after administration.
  Plasma samples were collected at different points for pharmacokinetic analysis.
CL/F | Measured on 1 hour before administration and 1, 2, 3, 4, 5, 6, 7, 8, 12, 24, 72, 96, 144, 192 hours after administration.
  Plasma samples were collected at different points for pharmacokinetic analysis.
Vz/F | Measured on 1 hour before administration and 1, 2, 3, 4, 5, 6, 7, 8, 12, 24, 72, 96, 144, 192 hours after administration.
  Plasma samples were collected at different points for pharmacokinetic analysis.
AUC0-∞ | Measured on 1 hour before administration and 1, 2, 3, 4, 5, 6, 7, 8, 12, 24, 72, 96, 144, 192 hours after administration.
  Plasma samples were collected at different points for pharmacokinetic analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, China, Wuhan, Hubei.China, China